CLINICAL TRIAL: NCT02341287
Title: Temperature Manipulating Gloves for the Treatment of Insomnia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in staffing and budget due to Covid-19
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Parker Hannifin Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1301013445
Record Dates: First submitted 2014-12-18; First posted 2015-01-19 (Estimated); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Warming hydrogel glove, then non-thermal glove (Active Comparator): In the first two-week period, subjects will wear a warming hydrogel glove. In the second two-week period, subjects will wear a non-thermal glove. Also a actigraph to monitor sleep latency.
  Interventions: Device: Warming hydrogel glove; Device: Non-thermal glove
- Non-thermal glove, then warming hydrogel glove (Placebo Comparator): In the first two-week period, subjects will wear a non-thermal glove. In the second two-week period, subjects will wear a warming hydrogel glove. Also an actigraph to monitor sleep latency.
  Interventions: Device: Warming hydrogel glove; Device: Non-thermal glove

INTERVENTIONS:
Device: Warming hydrogel glove — Subjects wore the warming hydrogel glove in either the first or second two-week period.
Device: Non-thermal glove — Subjects wore the non-thermal glove in either the first or second two-week period.

SUMMARY:
The investigators plan to test the effectiveness of warm gel gloves in reducing the time it takes individuals to fall asleep (sleep latency). The investigators will have subjects track their sleep for two-weeks using both sleep logs and a small wristwatch-like monitor called an actigraph to measure the degree of the persons' difficulty falling asleep. It must take at least 30-minutes to fall asleep 3-days per week to qualify for the study. If a subject qualifies, they will wear the heated gel gloves or a placebo non-heated gel glove during sleep for two-weeks and sleep will be measured again using sleep logs and actigraphy. The baseline sleep latency data will be compared to the treatment period using a independent t-test. The investigators believe that wearing the warm gel gloves will reduce sleep latency.

DETAILED DESCRIPTION:
Insomnia affects anywhere from six percent to 33% of the U.S. population depending on the precision of the definition being used. Therefore, represents one of the most prevalent health concerns for Americans. Individuals with insomnia frequently report problems such as (but not limited to) difficulty focusing and concentrating, memory difficulties, impaired motor coordination, irritability and impaired social interactions. Moreover, chronic insomnia has also been associated with reduced quality of life, higher absenteeism, impaired job performance, and higher healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for each participant are as follows: Must be between 18 and 65 years old
* Have difficulty initiating sleep for at least two-weeks, including a sleep latency of at least 30-minutes, three days per week (as measured by wrist actigraphy and/or sleep logs)
* No history of a dermatological disorders or chronic pain conditions
* Not currently using narcotics, psychotropic or hypnotic medications and willing to refrain from using these medications during the course of the study
* Limits caffeine consumption to less than or equal to 2 coffee servings, or equivalent per day
* Limits alcohol intake to 7-drinks per week and less than or equal to 1 drinks on any one night, must adjust alcohol consumption to 7-drinks per week and less than or equal to 1 drink on any one night for at least two weeks before study begins, and must not consume alcohol later than 8pm
* Naps less than or equal to 1-hour per week according to subjective report
* Must have a body mass index less than 30
* Shift workers will not be accepted.

Exclusion Criteria:

* History of a dermatological disorder
* Using narcotics, psychotropic or hypnotic medications
* Caffeine consumption greater than 2 coffee servings, or equivalent per day
* Alcohol intake greater than 7 drinks per week and greater than 1 drink on any one night, consume alcohol later than 8pm
* Naps greater than 1-hour per week according to subjective report
* Body mass index greater than 30; Shift worker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04-07 (Actual); Study Completion 2016-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ebben, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College Center for Sleep, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study utilizes a crossover design. Therefore, each subject is in both control and treatment groups.
Period: 1st Intervention (2 Weeks)
Arm/Group | Non-thermal Glove, Then Warming Hydrogel Glove | Warming Hydrogel Glove, Then Non-thermal Glove
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: 2nd Intervention (2 Weeks)
Arm/Group | Non-thermal Glove, Then Warming Hydrogel Glove | Warming Hydrogel Glove, Then Non-thermal Glove
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-thermal Glove, Then Warming Hydrogel Glove: In the first two-week period, subjects will wear a non-thermal glove. In the second two-week period, subjects will wear a warming hydrogel glove.
- Warming Hydrogel Glove, Then Non-thermal Glove: In the first two-week period, subjects will wear a warming hydrogel glove. In the second two-week period, subjects will wear a non-thermal glove.
- Total: Total of all reporting groups
Arm/Group | Non-thermal Glove, Then Warming Hydrogel Glove | Warming Hydrogel Glove, Then Non-thermal Glove | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency Assessed Via Actigraphy Monitoring
Description: The Outcome Measure will be assessed via actigraphy monitoring. Sleep latency will be measured on the actigraphy monitoring device and measured twice; during a two-week control period (non-thermal glove) and during the two-week treatment period (thermal hydrogel glove).
Time Frame: 2 weeks for each condition
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Non-thermal Glove | Warming Hydrogel Glove
Number analyzed (Participants) | 13 | 13
Minutes | 58.40 (25.29) | 44.39 (21.23)
Statistical Analysis 1: Comparison: Non-thermal Glove vs Warming Hydrogel Glove; Test type: Superiority; p = .023, t-test, 2 sided — Paired t-test of control average sleep latency vs. heated glove average sleep latency as measured by actigraph; Mean Difference (Net) = 14.01, 95% CI 2-sided [2.29 to 25.74], Standard Deviation 19.40

2. Secondary Outcome: Sleep Latency Assessed Via Sleep Log.
Description: Sleep latency measured in minutes via subjective sleep log.
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Non-thermal Glove | Warming Hydrogel Glove
Number analyzed (Participants) | 13 | 13
Minutes | 56.36 (23.56) | 42.84 (23.60)
Statistical Analysis 1: Comparison: Non-thermal Glove vs Warming Hydrogel Glove; Test type: Superiority — Paired t-test of control average sleep latency vs. heated glove average sleep latency as measured by sleep log; p < 0.014, t-test, 2 sided; Mean Difference (Net) = 13.51, 95% CI 2-sided [3.29 to 23.73], Standard Deviation 16.91

ADVERSE EVENTS:
Time Frame: 5-weeks
Groups:
- Non-thermal Glove: Subject received the non-thermal glove in either the first or second 2-week period of the study.
- Warming Hydrogel Glove: Subject received the warming hydrogel glove in either the first or second 2-week period of the study.
Arm/Group | Non-thermal Glove | Warming Hydrogel Glove
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No